CLINICAL TRIAL: NCT02295878
Title: Seaweed Derived Anti-inflammatory Agents and Antioxidants
Brief Title: The Effect of Seaweed Derived Polyphenols on Inflammation and Oxidative Stress in Vivo - The SWAFAX Study
Acronym: SWAFAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University of Reading (Other)
Responsible Party: Principal Investigator, Chris gill, Senior Lecturer, University of Ulster
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: REC/11/0077
Record Dates: First submitted 2014-11-03; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): 400mg capsule containing seaweed extract (treatment)
  Interventions: Dietary Supplement: Treatment capsule containing seaweed extract (treatment)
- Placebo (Placebo Comparator): 400mg capsule containing maltodextrin (placebo)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Treatment capsule containing seaweed extract (treatment) — 400mg capsule containing seaweed extract (treatment)
  Arms: Treatment
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Cardiovascular disease (CVD) is currently the leading cause of death worldwide. Epidemiologic studies have shown a diet rich in plant food protects against chronic degenerative diseases especially cardiovascular disease. Many of these studies have highlighted a potential role for phenolic compounds, which are abundant secondary plant metabolites, and which provide antioxidant and anti-inflammatory properties and are increasingly being shown to have an important role in influencing critical cell signalling pathways. A less well known, but nevertheless rich source of polyphenolic compounds is seaweed. In Ascophyllum nodosum, a common brown alga in the British Isles, polyphenols have been reported to comprise up to 14% of the dry weight of the plant. Some studies suggest that the potential antioxidant and anti-inflammatory benefits of seaweed-derived polyphenols may yield highly bioactive components with commercial potential for food and pharma applications. Preliminary work in our laboratory has revealed potent antioxidant activity of Ascophyllum nodosum extracts.

Therefore, the aim of this randomised, double-blind, placebo controlled, crossover design study is to investigate the biological activity of a food grade seaweed polyphenol extract in terms of reducing oxidative damage to DNA, modulation of inflammatory responses and reduction on chronic, low level inflammation in vivo. Apparently healthy volunteers (aged 30-65 years) will be randomised to receive either a capsule containing 100mg seaweed extract or a matched placebo daily for an 8 week period, with an 8 week washout period between each treatment. Fasting blood and urine samples will be taken from each volunteer at 4 time-points during the study, at baseline and completion of the 2 treatment phases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoker
* Omnivores and vegetarians
* Aged 30-65 years
* BMI >25kg/m2

Exclusion Criteria:

* Smokers
* Pregnant/lactating women
* Vegans
* Diabetes mellitus, CVD
* Autoimmune/inflammatory disorders
* History of neoplasm
* Recent acute illness
* Anti-inflammatory medication
* Habitual use of vitamin supplements

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
DNA damage in lymphocytes (Comet assay) | 8 weeks
  To assess the DNA damage in lymphocytes using the Comet assay

SECONDARY OUTCOMES:
Intracellular cytokine analysis (Tissue Factor expression using flow cytometry) | 8 weeks
  To assess intracellular cytokine levels in lymphocyte and monocyte populations and Tissue Factor expression using flow cytometry

OTHER OUTCOMES:
C-reactive protein | 8 weeks
  C-reactive protein measured on an iLAB 600 analyser
Oxidative stress using isoprostanes | 8 weeks
  Oxidative stress will be assessed using isoprostanes
Total cholesterol | 8 weeks
  Total cholesterol measured in plasma on an iLAB 600 analyser
HDL cholesterol | 8 weeks
  HDL cholesterol measured in plasma on an iLAB 600 analyser
Triglycerides | 8 weeks
  Triglycerides measured in plasma on an iLAB 600 analyser

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gill, BSc, PhD, Principal Investigator — Ulster University

REFERENCES:
- [Derived] Baldrick FR, McFadden K, Ibars M, Sung C, Moffatt T, Megarry K, Thomas K, Mitchell P, Wallace JMW, Pourshahidi LK, Ternan NG, Corona G, Spencer J, Yaqoob P, Hotchkiss S, Campbell R, Moreno-Rojas JM, Cuevas FJ, Pereira-Caro G, Rowland I, Gill CIR. Impact of a (poly)phenol-rich extract from the brown algae Ascophyllum nodosum on DNA damage and antioxidant activity in an overweight or obese population: a randomized controlled trial. Am J Clin Nutr. 2018 Oct 1;108(4):688-700. doi: 10.1093/ajcn/nqy147. PMID 30321272